CLINICAL TRIAL: NCT01765738
Title: Randomized Double Blind Comparison of an Antibiotic Impregnated PICC Catheter Versus a Regular PICC Catheter in a Tertiary Care Setting
Brief Title: Comparison of an Antibiotic Impregnated PICC Catheter Versus a Regular PICC Catheter in a Tertiary Care Setting
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Project never received funding.
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PICC Line Comparison
Record Dates: First submitted 2013-01-08; First posted 2013-01-10 (Estimated); Last update posted 2018-06-18 (Actual); Status verified 2016-09

CONDITIONS: Peripherally Inserted Central Catheters
Keywords: PICC
MeSH Terms: interventions — Catheterization, Peripheral

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antibiotic coated PICC (Active Comparator): Cook Medical Spectrum Turbo-Ject Minocycline/Rifampin Power-Injectable PICC (5fr double lumen or 6fr triple lumen)
  Interventions: Device: PICC (Cook, Bard)
- Non-antibiotic coated PICC (Active Comparator): Bard Access PowerPICC Power Injection PICCs (6fr double lumen or 6fr. triple lumen)
  Interventions: Device: PICC (Cook, Bard)

INTERVENTIONS:
Device: PICC (Cook, Bard) — Comparison of antibiotic coated PICC vs. non-coated PICC
  Other Names: Minocycline/Rifampin Power-Injectable PICC; PowerPICC Power Injection PICCs

SUMMARY:
To determine whether antibiotic impregnated PICC catheters have a lower infection rate than a conventional PICC catheter in a tertiary care patient population. Secondary goals will be to determine if there is a difference between the two catheters with early and late infections, to determine the cost comparison including extra cost of treatment for a line related infection, to determine if there are any non-infectious related complication differences between the two catheters.

DETAILED DESCRIPTION:
All patients who are referred to VIR for a PICC line will be evaluated to see if they satisfy the inclusion/exclusion criteria. The study will be discussed with those who do and informed consent will be obtained from those wishing to participate. The patient will then be randomized to one of two types of PICC lines. All lines will be placed by identical technique. This will include sterile technique, placement via a vein of the upper arm using ultrasound guidance, and positioning of the catheter tip under fluoroscopic guidance. A database of all catheters placed will be kept. Records will be reviewed at 1 week, 30 days, and 60 days by the Interventional Radiology Fellow.Review will include length of time catheter was in place, whether treatment was completed, whether catheter was removed prematurely, the clinical reason for removal, results of other imaging tests, and results of cultures on any catheters removed for suspicion of infection. Any non-infectious complications related to the catheter will also be noted. The reviewer will be blinded to which catheter was used during the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 18 years of age
* Have been scheduled for a medically necessary PICC placement

Exclusion Criteria:

* Less than 18 years of age

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-02; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Infection rate | 60 days
  Records will be reviewed up to 60 days post PICC line procedure to assess whether catheter was removed prematurely for infection and results of cultures on any catheters removed.

CONTACTS AND LOCATIONS:
Overall Officials: J. Bayne Selby, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States